CLINICAL TRIAL: NCT03387956
Title: Intravenous Dexamethasone Combined With Intrathecal Atropine to Prevent Morphine-related Nausea and Vomiting After Cesarean Delivery: A Randomized Double-blinded Study
Brief Title: Intrathecal Atropine to Prevent Postoperative Nausea and Vomiting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Emad Zarief , MD, Dr, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00009916
Record Dates: First submitted 2017-12-20; First posted 2018-01-02 (Actual); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Postoperative Nausea
Keywords: Postoperative Nuasea
MeSH Terms: conditions — Postoperative Nausea and Vomiting | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Atropine group (Active Comparator): Atropine group (A): Patients received intrathecal heavy Marcaine, 2 ml, 0.5% plus 300 µg morphine and 100 µg atropine (0.5ml), and intravenous injection of 2ml normal saline.
  Interventions: Drug: Intrathecal atropine
- Dexamethasone group (Active Comparator): Dexamethasone group (D): Patients received intrathecal heavy Marcaine 2 ml, 0.5% plus 300 µg morphine (0.5ml), and intravenous 8 mg dexamethasone (2ml).
  Interventions: Drug: dexamethasone
- Dexamethasone and Atropine group (Active Comparator): Dexamethasone and Atropine group (DA): Patients received intrathecally as group A, plus intravenous injection of 2 ml, dexamethasone 8 mg. Postoperative follow-up of both nausea and vomiting was done over 24 hours postoperative.
  Interventions: Drug: Intrathecal atropine; Drug: dexamethasone

INTERVENTIONS:
Drug: Intrathecal atropine — 100ug intrathecal atropine will be injected with spinal anesthesia
  Arms: Atropine group; Dexamethasone and Atropine group
Drug: dexamethasone — intravenous 8 mg dexamethasone (2ml).
  Arms: Dexamethasone and Atropine group; Dexamethasone group

SUMMARY:
optimal postoperative pain control with intrathecal morphine, with proper prevention of postoperative nausea and vomiting. Dexamethasone, and or atropine could offer some protection against nausea and vomiting.

DETAILED DESCRIPTION:
One of the gold standards for analgesia following cesarean delivery is intrathecal morphine, which is not devoid of complications namely postoperative nausea and vomiting. We evaluated the antiemetic effect of intravenous dexamethasone combined with intrathecal atropine after cesarean delivery under spinal bupivacaine plus morphine anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* females
* 18-40 years of age
* elective cesarean delivery under bupivacaine spinal anesthesia

Exclusion Criteria:

* renal disease
* preeclampsia
* liver disease
* cardiac disease
* Coagulopathy
* chronic cough
* nausea
* vomiting
* patient refusal

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2017-03-20 (Actual); Primary Completion 2017-07-28 (Actual); Study Completion 2017-08-10 (Actual)

PRIMARY OUTCOMES:
postoperative nausea | 24 hours
  Monitoring scale of nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Emad Zarief Kamel Said, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided